CLINICAL TRIAL: NCT04264442
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, 48-Week, Parallel-Group Study of the Efficacy and Safety of Losmapimod in Treating Subjects With Facioscapulohumeral Muscular Dystrophy (FSHD) With Open-Label Extension (OLE)
Brief Title: Efficacy and Safety of Losmapimod in Treating Subjects With Facioscapulohumeral Muscular Dystrophy (FSHD) With Open-Label Extension (OLE)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Fulcrum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIS-002-2019 OLE
Record Dates: First submitted 2020-01-30; First posted 2020-02-11 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Facioscapulohumeral Muscular Dystrophy (FSHD)
Keywords: FSHD, FSHD1; Muscular Dystrophy; Muscular Dystrophies; Facioscapulohumeral Muscular Disorders; Musculoskeletal Diseases; Neuromuscular Diseases
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies; Musculoskeletal Diseases; Neuromuscular Diseases | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Intervention Model Description: This study is part two of NCT04003974 which was a randomized, double-blind placebo-controlled treatment period for 48 weeks. This study is an open-label extension with losmapimod in patients with FSHD1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Losmapimod (Experimental): FSHD1 patients with genetic confirmation will receive Losmapimod 15 mg by mouth twice daily for a total of 30 mg daily until 90 days after commercial drug is available post regulatory approval or until the study is discontinued by the Sponsor.
  Interventions: Drug: Losmapimod

INTERVENTIONS:
Drug: Losmapimod — Patients will receive Losmapimod 15 mg by mouth twice daily for a total of 30 mg daily until 90 days after commercial drug is available post regulatory approval or until the study is discontinued by the Sponsor. The study drug should be taken with food and the date and time of each dose taken should be recorded in the subject diary.

SUMMARY:
This study is an open-label extension to evaluate the safety and tolerability of long-term dosing of Losmapimod in patients with FSHD1 who participated in the ReDux4 study.

DETAILED DESCRIPTION:
This study is an open-label extension study to evaluate the safety and tolerability of long-term dosing of Losmapimod in patients with FSHD1 who participated in the ReDux4 study.

This study is a multi-center clinical trial. It will be conducted in North America, Canada and Europe. Only patients who participated and competed all study procedures in the ReDUX4 Study treatment period will be eligible to participate in this open label extension study.

Patients who complete the randomized, placebo-controlled portion of the study will have the option to roll over into the open-label extension study.

Patients will receive 15 mg of losmapimod by mouth twice daily for a total of 30 mg by mouth daily. All patients will attend clinic visits approximately every 12 weeks.

Participation in this open-label extension study will continue until 90 days after losmapimod becomes commercially available, the patient withdraws from the study, or the Sponsor decides to close the study.

The primary endpoint of the study is to evaluate the safety and tolerability of long-term dosing of losmapimod in patients with FSHD.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have consented to participate and must have provided signed, dated and witnessed an IRB-approved informed consent form that conforms to federal and institutional guidelines.
* Male or female subjects
* Patients must be between 18 and 65 years of age, inclusive
* Must be willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines and other study procedures.
* Will practice an approved method of birth control

Exclusion Criteria:

* Has a history of any illness or any clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject. This may include, but is not limited to, a history of relevant drug or food allergies; history of cardiovascular or central nervous system disease; neuromuscular diseases except FSHD (eg, myopathy, neuropathy, neuromuscular junction disorders); or clinically significant history of mental disease.
* For subjects who are on drug(s) or supplements that may affect muscle function, as determined by the treating physician, or that are included in the list of drugs presented in the protocol, subjects must be on a stable dose of that drug(s) or supplement for at least 3 months prior to the first dose of study drug and remain on that stable dose for the duration of the study. Changes to the dose or treatment discontinuation during the study can only be done for strict medical reasons by the treating physician with clear documentation and notification to the sponsor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Helene Jouvin, MD, Study Director — Fulcrum Therapeutics
Locations (17):
- United States (12):
  - University of California Irvine, Irvine, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State University, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washinton Medical Center, Seattle, Washington
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- CHU de NICE- CHU pasteur2, Nice, France
- Spain (2):
  - Hospital de la Sta Creu i St Pau, Barcelona
  - Hospital UiP La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbour AM, Sarov-Blat L, Cai G, Fossler MJ, Sprecher DL, Graggaber J, McGeoch AT, Maison J, Cheriyan J. Safety, tolerability, pharmacokinetics and pharmacodynamics of losmapimod following a single intravenous or oral dose in healthy volunteers. Br J Clin Pharmacol. 2013 Jul;76(1):99-106. doi: 10.1111/bcp.12063. PMID 23215699
- [Background] Cheriyan J, Webb AJ, Sarov-Blat L, Elkhawad M, Wallace SM, Maki-Petaja KM, Collier DJ, Morgan J, Fang Z, Willette RN, Lepore JJ, Cockcroft JR, Sprecher DL, Wilkinson IB. Inhibition of p38 mitogen-activated protein kinase improves nitric oxide-mediated vasodilatation and reduces inflammation in hypercholesterolemia. Circulation. 2011 Feb 8;123(5):515-23. doi: 10.1161/CIRCULATIONAHA.110.971986. Epub 2011 Jan 24. PMID 21262998
- [Background] de Greef JC, Lemmers RJ, van Engelen BG, Sacconi S, Venance SL, Frants RR, Tawil R, van der Maarel SM. Common epigenetic changes of D4Z4 in contraction-dependent and contraction-independent FSHD. Hum Mutat. 2009 Oct;30(10):1449-59. doi: 10.1002/humu.21091. PMID 19728363
- [Background] Han JJ, Kurillo G, Abresch RT, de Bie E, Nicorici A, Bajcsy R. Reachable workspace in facioscapulohumeral muscular dystrophy (FSHD) by Kinect. Muscle Nerve. 2015 Feb;51(2):168-75. doi: 10.1002/mus.24287. Epub 2014 Nov 19. PMID 24828906
- [Background] Jagannathan S, Shadle SC, Resnick R, Snider L, Tawil RN, van der Maarel SM, Bradley RK, Tapscott SJ. Model systems of DUX4 expression recapitulate the transcriptional profile of FSHD cells. Hum Mol Genet. 2016 Oct 15;25(20):4419-4431. doi: 10.1093/hmg/ddw271. PMID 28171552
- [Background] Statland JM, Tawil R. Risk of functional impairment in Facioscapulohumeral muscular dystrophy. Muscle Nerve. 2014 Apr;49(4):520-7. doi: 10.1002/mus.23949. Epub 2014 Feb 10. PMID 23873337
- [Background] Wang LH, Friedman SD, Shaw D, Snider L, Wong CJ, Budech CB, Poliachik SL, Gove NE, Lewis LM, Campbell AE, Lemmers RJFL, Maarel SM, Tapscott SJ, Tawil RN. MRI-informed muscle biopsies correlate MRI with pathology and DUX4 target gene expression in FSHD. Hum Mol Genet. 2019 Feb 1;28(3):476-486. doi: 10.1093/hmg/ddy364. PMID 30312408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed either 24 or 48 weeks in the placebo-controlled treatment period of the parent study were eligible to enroll in the Open-Label Extension (OLE) phase. A total 76 participants entered the OLE) phase and received at least 1 dose of losmapimod. Of those, 39 were previously in the losmapimod group and 37 in the placebo group during the double-blind treatment period of study (NCT04003974) and met eligibility criteria for continued treatment.
Pre-assignment Details: Participants were analysed according to their original treatment assignment and their entry point into the OLE: Losmapimod 15 mg BID / Losmapimod 15 mg BID (from Week 24 or Week 48) and Placebo BID / Losmapimod 15 mg BID (from Week 24 or Week 48).
Groups:
- Losmapimod 15 Milligrams (mg) Twice Daily (BID): Participants will continue to receive Losmapimod 15 mg (2×7.5 mg tablets/dose) BID until 90 days after commercial drug is available post regulatory approval or until the study is discontinued by the Sponsor (up to 60 months).
Period: Overall Study
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Started | 76
Completed | 29
Not Completed | 47
Not completed — Lack of Efficacy | 6
Not completed — Lost to Follow-up | 2
Not completed — Sponsor Decision | 23
Not completed — Withdrawal by Subject | 11
Not completed — Study Termination | 5

BASELINE CHARACTERISTICS:
Population: Open-Label Analysis Set comprised of all participants who completed 24 or 48 weeks of treatment in the placebo-controlled treatment period and received at least 1 dose of open-label losmapimod in the OLE.
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.2 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 69
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 66
  More than one race | 1
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Serious Treatment Emergent Adverse Events (Serious TEAEs) and TEAEs
Description: A TEAE is an adverse event that begins on or after the first dose of study drug and on or before the stop of study drug plus 7 days or begins before the first dose of study drug and worsens on or after the first dose of study drug and on or before the stop of study drug plus 7 days. An adverse event with completely missing onset and end dates was considered as TEAE. An adverse event with missing onset date but the end date is on or after the first dose of study drug and before the stop of study drug plus 7 days was considered a TEAE.
Time Frame: Up to 57 months
Population: Open-Label Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 76
Participants
  Any serious TEAE | 7
  Any TEAE | 71

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Chemistry Parameters
Description: Blood samples were collected for the analysis of chemistry parameters: Glucose, sodium, potassium, calcium, inorganic phosphate, total protein, albumin, blood urea nitrogen, creatinine, total bilirubin, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase and creatine phosphokinase.
Time Frame: Up to 57 months
Population: Open-Label Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 76
Participants | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: Blood samples were collected for the analysis of hematology parameters: hemoglobin (including mean corpuscular volume), mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, hematocrit, red blood cell count, total white blood cell count, platelet count. Differential blood counts, including basophils, eosinophils, neutrophils, lymphocytes, and monocytes
Time Frame: Up to 57 months
Population: Open-Label Analysis Set:
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 76
Participants | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Serum Coagulation Parameters
Description: Blood samples were collected for the analysis of Serum coagulation parameters: International normalized ratio, prothrombin time, partial thromboplastin time.
Time Frame: Up to 57 months
Population: Open-Label Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 76
Participants | 0

5. Primary Outcome: Number of Participants With Clinically Significant Changes in Urinalysis
Description: Urine samples were collected for the analysis of urinalysis parameters: Leucocytes, blood, nitrite, protein, urobilinogen, bilirubin, pH, specific gravity, ketones, glucose.
Time Frame: Up to 57 months
Population: Open-Label Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 76
Participants | 0

6. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Parameters
Description: Vital parameters including pulse rate, respiration rate, blood pressure, and temperature were measured in seated or recumbent for at least 5 minutes. Data for number of participants with abnormal clinically significant changes for vital signs have been presented.
Time Frame: Up to 57 months
Population: Open-Label Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 76
Participants | 0

7. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Parameters
Description: Twelve-lead ECGs was performed after participants has been recumbent for at least 5 minutes.
Time Frame: Up to 57 months
Population: Open-Label Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 76
Participants | 0

8. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examinations
Description: Physical examinations included an evaluation of body systems, including but not limited to the following: skin; head, eyes, ears, nose, and throat; respiratory system; cardiovascular system; abdomen (liver, spleen); lymph nodes; neurological system; and musculoskeletal system.
Time Frame: Up to 57 months
Population: Open-Label Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 76
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 57 months
Description: Serious TEAEs and TEAEs were collected in Open-Label Analysis Set which comprised of all participants who completed 24 or 48 weeks of treatment in the placebo-controlled treatment period and received at least 1 dose of open-label losmapimod in the OLE.
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
All-Cause Mortality (participants affected / at risk) | 0/76
Serious Adverse Events (participants affected / at risk) | 7/76
Other Adverse Events (participants affected / at risk) | 71/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Losmapimod 15 Milligrams (mg) Twice Daily (BID) (N=76)
Acute myocardial infarction (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 1
Ulcer haemorrhage (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 1
Labile blood pressure (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Losmapimod 15 Milligrams (mg) Twice Daily (BID) (N=76)
Palpitations (Cardiac disorders) | 4
Dry eye (Eye disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 4
Food poisoning (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 8
Pain (General disorders) | 4
Corona virus infection (Infections and infestations) | 37
Influenza (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 15
Sinusitis (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 8
Arthropod bite (Injury, poisoning and procedural complications) | 4
Contusion (Injury, poisoning and procedural complications) | 11
Fall (Injury, poisoning and procedural complications) | 28
Joint injury (Injury, poisoning and procedural complications) | 4
Ligament sprain (Injury, poisoning and procedural complications) | 6
Skin abrasion (Injury, poisoning and procedural complications) | 5
Skin laceration (Injury, poisoning and procedural complications) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Headache (Nervous system disorders) | 9
Anxiety (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 5
Nephrolithiasis (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT04264442/Prot_002.pdf
  • Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT04264442/SAP_001.pdf